CLINICAL TRIAL: NCT00488826
Title: An Open-Label Controlled Phase I/III Study to Evaluate the Safety and Immunogenicity of Pneumococcal 7-Valent Conjugate Vaccine [DIPHTHERIA CRM197 PROTEIN] (PrevenarTM) in Healthy Infants
Brief Title: Study Evaluating 7-Valent Pneumococcal Conjugate Vaccine in Healthy Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0887X-101518
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2009-05-27 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Pneumococcal Infections
Keywords: Vaccines, Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Tetanus Toxoid

INTERVENTIONS:
Biological: 7-valent pneumococcal conjugate vaccine
Biological: Diptheria and tetanus toxoids and accelular pertussis vaccine (DTaP)

SUMMARY:
This study is a combination of a Phase I and Phase III study design. The Phase I portion is an open-label, controlled study to evaluate the safety of 7vPnC in healthy Chinese infants. The Phase III portion is an open-label, controlled, randomized study to evaluate the safety and immunogenicity of 7-Valent Pneumococcal Conjugate Vaccine (7vPnC)in healthy Chinese infants. Both phases include a Primary Series which includes the primary 3 doses of 7vPnC and /or Diptheria and tetanus toxoids and accelular pertussis vaccine (DTaP) at about 3, 4, and 5 months of age; and a Booster Dose which includes the 4th dose of 7vPnC at 12-15 months of age.

DETAILED DESCRIPTION:
This study is a combination of a Phase I and Phase III study design. The Phase I portion is an open-label, controlled study to evaluate the safety of 7vPnC in healthy Chinese infants. The Phase III portion is an open-label, controlled, randomized study to evaluate the safety and immunogenicity of 7vPnC in healthy Chinese infants. Both phases include a Primary Series which includes the primary 3 doses of 7vPnC and/or DTaP at about 3, 4, and 5 months of age; and a Booster Dose which includes the 4th dose of 7vPnC at 12-15 months of age. A total of 822 healthy Chinese infants will be enrolled. The study will be conducted in 2 phases: Phase I and Phase III.

Phase I: 22 healthy infants will be enrolled first and receive a dose of 7vPnC at least 7 days prior to receiving DTaP and followed up on safety for 30 days post the immunization. If there are no adverse events of specific concern considered, in the opinion of the principal investigator, related to the study vaccine (including, though not limited to, infectious and allergic reactions as described in the China Immunization Handbook) within 4 days after the first dose immunization and no serious adverse event possibly, probably or definitely related to the study vaccine within 30 days after the first dose of immunization, Phase III can be initiated and the infants in Phase I will proceed to the next dose of the Primary Series. If such events occur, a medical review will be conducted by both the investigator and the Sponsor to decide if the study can proceed.

Phase III: 800 infants will be enrolled and randomized to one of 3 groups according to the administration regimen. Group 1: 300 infants will receive the primary 3 doses of 7vPnC separately at 3, 4 and 5 months of age. Group 2: 300 infants will receive the primary 3 doses of 7vPnC concurrently with DTaP at 3, 4 and 5 months of age. Group 3: 200 infants will receive DTaP only at 3, 4 and 5 months of age. The injection site is the left upper arm deltoid for 7vPnC and the right upper arm deltoid for DTaP.

Safety Evaluation: Each infant will have an initial physical examination and history obtained at the enrollment visit and a brief physical evaluation at each subsequent visit. Following immunization, each subject will be observed in the clinic for 30 minutes and evaluated for signs or symptoms of anaphylaxis and reactions at the injection sites. The parent or legal guardian will be required to take the infant's axillary temperature on the evening of immunization and for 3 consecutive evenings following the immunization. In addition, if the parent suspects that the infant may have a fever at any time in the four days following immunization, the temperature is to be taken and recorded. Thermometers for axillary temperature use and diary cards will be supplied by Wyeth for distribution to the parents.

The parent or legal guardian of each subject will be instructed to complete a diary card for 4 days [day of immunization (day 0) and next 3 days] following each immunization. Information collected will include: the subject's axillary temperature, local reactions at the 7vPnC injection site (All subjects in Phase I of the study and Group 1 and Group 2 of Phase III) and DTaP injection site (Group 2 and Group 3 of Phase III) (tenderness, presence and size of erythema and induration/swelling) and any systemic reactions (disrupted sleep, drowsiness, decreased appetite, irritability, vomiting, diarrhea and rash not limited to the injection site) occurring days 0-3. The subject will return to clinic or be visited at home on the day after immunization (Day 1) for local and systemic reaction observation by study personnel. The parent or legal guardian will be contacted by telephone or home visit at 2 and 3 days post-immunization to collect information on local and systemic events and the information will be recorded on the source data sheet by study personnel. On, or after, the fourth day after each immunization, the study personnel will collect the diary card. The data in the diary card will be reconciled with the data in the source data sheet. If there is discrepancy, it should be clarified with the parents and recorded.

At the visit of next immunization, the interim medical history since Day 4 post last immunization will be reviewed with the parent/legal guardian. If there is any adverse event, it should be collected and recorded in the case report form. The primary source of data on adverse events will be the parent or legal guardian of each subject, as well as any medical records from a health care provider sought as a result of an adverse event. The parent/legal guardian is instructed to contact the investigators immediately for any serious adverse events.

Assessment of Immunogenicity: Up to 3ml venous blood will be collected from 55 infants in Group 1, 55 infants in Group 2 and 55 infants in Group 3 of Phase III, immediately prior to the first dose and 30-40 days after the 3rd dose to assess the immunogenicity.

Booster Dose: All infants in Phase I and Group 1 and Group 2 of Phase III will receive the booster dose of 7vPnC at 12-15 months of age. Local/systemic reactions will be observed in the same way as after the primary dose.

Assessment of Immunogenicity: Up to 3ml venous blood will be collected from the same 55 infants in Group 1 and 55 infants in Group 2 as in the Primary Series of Phase III, immediately prior to the forth dose and 30-40 days after the 4th dose to assess the immunogenicity.

The statistical analysis of the two phases will be conducted separately. The statistical analysis of the primary series is planned when all subjects have received the 1st, 2nd and 3rd dose of 7vPnC and 3 doses of DTaP or 3 doses of DTaP alone and the 30-day safety follow-up period has terminated. The analysis of the booster dose is planned when all subjects have received the 4th dose of 7vPnC and the 30-day safety follow-up period has terminated.

ELIGIBILITY:
Inclusion Criteria:

* Chinese infants, aged 3-4 months (90-120 days) at enrollment, and have not received their 1st dose of DTaP
* In good health determined by medical history, physical examination (axillary temperature and weight) and clinical judgment of the investigator
* An informed consent form must be signed by at least one of the parent/legal guardian. The parent or legal guardian are willing to adhere to the regimen of the study and are capable of using the thermometer, calipers and filling out the diary card

Exclusion Criteria:'

* Weight < 2 SD for age
* History of neurological disorders including a personal and family history of convulsion and epilepsy (including febrile seizures)
* Receipt of blood products, including gamma globulin within 12 weeks prior to study entry
* Hypersensitivity to any component of 7vPnC, including diphtheria toxoid
* Known previous anaphylactic reactions to any vaccines or medicines
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection
* Known or suspected impairment of immune function due to the use of immunosuppressive therapy (including irradiation, corticosteroids, antimetabolites, alkylating agents, and cytotoxic agents), a genetic defect, HIV infection or other cause
* History of culture-proven invasive disease caused by S. pneumoniae
* Any significant congenital deformity or serious chronic diseases
* Previous immunization with licensed or investigational pneumococcal vaccine
* Other investigational medicine is being administered or has been administered within 12 weeks before screening or participation in another investigational study

Ages: 90 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2005-10; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in China from September 2006 to May 2007.
Pre-assignment Details: Subjects were enrolled into study according to inclusion/exclusion criteria without a screening period.
Groups:
- 7vPnC Separately: 7-valent pneumococcal conjugate vaccine (7vPnC) administered at 3, 4, and 5 months of age. Diphtheria and tetanus toxoids and accelular pertussis vaccine (DTaP) administered at least 7 days after 7vPnC at 3, 4, and 5 months of age.
- 7vPnC + DTaP Concurrently: 7vPnC adminstered concurrently with DTaP at 3, 4, and 5 months of age.
- DTaP Alone: DTaP administered at 3, 4, and 5 months of age.
Period: Overall Study
Arm/Group | 7vPnC Separately | 7vPnC + DTaP Concurrently | DTaP Alone
Started | 300 | 296 | 204
Completed | 244 | 244 | 178
Not Completed | 56 | 52 | 26
Not completed — Withdrawal by Subject | 40 | 35 | 19
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Adverse Event | 9 | 15 | 4
Not completed — Lost to Follow-up | 5 | 1 | 0
Not completed — Protocol Deviations | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7vPnC Separately | 7vPnC + DTaP Concurrently | DTaP Alone | Total
Number analyzed (Participants) | 300 | 296 | 204 | 800
Age Continuous [Median (Standard Deviation); unit: months] | 3.5 (1.0) [3.0 to 4.0] | 3.5 (1.0) [3.0 to 4.0] | 3.5 (1.7) [3.0 to 4.7] | 3.5 (1.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 133 | 81 | 356
  Male | 158 | 163 | 123 | 444

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Serotype-Specific IgG Antibodies
Description: Vaccine efficacy can be assessed by measuring the levels of antibodies to the specific types (or serotypes) of bacteria covered by the vaccine. IgG antibodies for the 7 pneumococcal serotypes in 7vPnC (4, 6B, 9V, 14, 18C, 19F, 23F) were assessed 30-50 days after the third dose of vaccine. Antibody levels were measured by standardized enzyme-linked immunosorbent assay (ELISA). The minimum level of antibodies required to confer protection has been defined as 0.15 ug/ml by the Northern California Kaiser Permanente (NCKP) study, and as 0.35 ug/ml by the World Health Organization (WHO).
Time Frame: 7 months
Population: Population analyzed was available immunogenicity population (all subjects who completed the primary series of 7vPnC or DTaP and had the post-third dose serum available for assessment) and were in either the "7vPnC separately" or "DTaP alone" group. The "7vPnC + DTaP" group was not part of the primary objective; no statistical testing was done.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/ml
Arm/Group | 7vPnC Separately | 7vPnC + DTaP Concurrently | DTaP Alone
Number analyzed (Participants) | 64 | 0 | 47
ug/ml
  Serotype 4 | 15.26 [12.51 to 18.61] |  | 0.01 [0.01 to 0.02]
  Serotype 6B | 3.1 [2.15 to 4.46] |  | 0.06 [0.04 to 0.08]
  Serotype 9V | 6.82 [5.65 to 8.23] |  | 0.06 [0.05 to 0.09]
  Serotype 14 | 17.75 [13.53 to 23.28] |  | 0.14 [0.09 to 0.22]
  Serotype 18C | 6.24 [5.07 to 7.69] |  | 0.03 [0.02 to 0.04]
  Serotype 19F | 11.77 [8.91 to 15.54] |  | 0.07 [0.05 to 0.10]
  Serotype 23F | 4.7 [3.22 to 6.86] |  | 0.05 [0.03 to 0.08]
Statistical Analysis 1: Comparison: 7vPnC Separately vs DTaP Alone; The ratio of the "7vPnC Separately" group to the "DTaP Alone" group geometric mean comparisons (GMC) was provided with a corresponding 90% confidence interval; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 1097, 90% CI [793.6 to 1461] — This analysis is for Serotype 4
Statistical Analysis 2: Comparison: 7vPnC Separately vs DTaP Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 54.6, 90% CI [35.36 to 85.49] — This analysis is for Serotype 6B
Statistical Analysis 3: Comparison: 7vPnC Separately vs DTaP Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 99.48, 90% CI [79.81 to 142.0] — This analysis is for Serotype 9V
Statistical Analysis 4: Comparison: 7vPnC Separately vs DTaP Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 134.3, 90% CI [80.83 to 197.1] — This analysis is for Serotype 14
Statistical Analysis 5: Comparison: 7vPnC Separately vs DTaP Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 200.3, 90% CI [151.9 to 302.4] — This analysis is for Serotype 18C
Statistical Analysis 6: Comparison: 7vPnC Separately vs DTaP Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 181.3, 90% CI [119.8 to 253.1] — This analysis is for Serotype 19F
Statistical Analysis 7: Comparison: 7vPnC Separately vs DTaP Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 90.02, 90% CI [57.93 to 150.5] — This analysis is for Serotype 23F

2. Secondary Outcome: Concentration of Serotype-Specific IgG Antibodies
Description: Vaccine efficacy can be assessed by measuring the levels of antibodies to the specific types (or serotypes) of bacteria covered by the vaccine. IgG antibodies for the 7 pneumococcal serotypes in 7vPnC (4, 6B, 9V, 14, 18C, 19F, 23F) were assessed 30-50 days after the third dose of vaccine. Antibody levels were measured by standardized enzyme-linked immunosorbent assay (ELISA). The minimum level of antibodies required to confer protection has been defined as 0.15 ug/ml by the Northern California Kaiser Permanente (NCKP) study and as 0.35 ug/ml by the World Health Organization (WHO).
Time Frame: 7 months
Population: The population analyzed was all the available immunogenicity population (all subjects who completed the primary series of 7vPnC or DTaP and had the post third dose serum available for assessment) and were in either "7vPnC+DTaP Concurrently" or "DTaP Alone" group. The "7vPnC Separately" group was not included as part of this objective.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/ml
Arm/Group | 7vPnC Separately | 7vPnC + DTaP Concurrently | DTaP Alone
Number analyzed (Participants) | 0 | 66 | 47
ug/ml
  Serotype 4 |  | 8.99 [7.59 to 10.66] | 0.01 [0.01 to 0.02]
  Serotype 6B |  | 1.19 [0.86 to 1.64] | 0.06 [0.04 to 0.08]
  Serotype 9V |  | 4.9 [3.89 to 6.16] | 0.06 [0.05 to 0.09]
  Serotype 14 |  | 13.35 [10.31 to 17.29] | 0.14 [0.09 to 0.22]
  Serotype 18C |  | 4.77 [3.79 to 6.00] | 0.03 [0.02 to 0.04]
  Serotype 19F |  | 5.62 [4.45 to 7.09] | 0.07 [0.05 to 0.10]
  Serotype 23F |  | 2.27 [1.68 to 3.06] | 0.05 [0.03 to 0.08]
Statistical Analysis 1: Comparison: 7vPnC + DTaP Concurrently vs DTaP Alone; The ratio of the "7vPnC + DTaP Concurrently" group to "DTaP Alone" group geometric mean comparisons (GMC) was provided with a corresponding 90% confidence interval; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 665.1, 90% CI [473.3 to 851.2] — This analysis is for Serotype 4
Statistical Analysis 2: Comparison: 7vPnC + DTaP Concurrently vs DTaP Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 22.2, 90% CI [13.99 to 31.77] — This analysis is for Serotype 6B
Statistical Analysis 3: Comparison: 7vPnC + DTaP Concurrently vs DTaP Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 73.7, 90% CI [56.41 to 103.6] — This analysis is for Serotype 9V
Statistical Analysis 4: Comparison: 7vPnC + DTaP Concurrently vs DTaP Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 99.48, 90% CI [61.09 to 147.5] — This analysis is for Serotype 14
Statistical Analysis 5: Comparison: 7vPnC + DTaP Concurrently vs DTaP Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 164, 90% CI [114.9 to 232.9] — This analysis is for Serotype 18C
Statistical Analysis 6: Comparison: 7vPnC + DTaP Concurrently vs DTaP Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 81.45, 90% CI [57.98 to 119.1] — This analysis is for Serotype 19F
Statistical Analysis 7: Comparison: 7vPnC + DTaP Concurrently vs DTaP Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; P-Values were not calculated; Geometric mean ratio = 44.7, 90% CI [29.48 to 68.71] — This analysis is for Serotype 23F

ADVERSE EVENTS:
Arm/Group | 7vPnC Separately | 7vPnC + DTaP Concurrently | DTaP Alone
Serious Adverse Events (participants affected / at risk) | 3 | 7 | 1
Other Adverse Events (participants affected / at risk) | 206 | 263 | 137
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | 7vPnC Separately | 7vPnC + DTaP Concurrently | DTaP Alone
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 0/297 | 5/295 | 1/201
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1/297 | 2/295 | 0/201
Enteritis (Gastrointestinal disorders) | 1/297 | 1/295 | 1/201
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0/297 | 1/295 | 0/201
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1/297 | 0/295 | 0/201
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1/297 | 0/295 | 0/201
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | 7vPnC Separately | 7vPnC + DTaP Concurrently | DTaP Alone
Diarrhea (Gastrointestinal disorders) | 33/297 | 54/295 | 28/201
Pyrexia (General disorders) | 59/297 | 82/295 | 50/201
Nasopharyngitis (Infections and infestations) | 39/297 | 54/295 | 28/201
Upper respiratory tract infection (Infections and infestations) | 20/297 | 15/295 | 0/201
Cough (Respiratory, thoracic and mediastinal disorders) | 55/297 | 58/295 | 31/201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.